CLINICAL TRIAL: NCT07197515
Title: Legal Evaluation for Greater Access to Cancer Care (LEGAL-CARE): A Pilot Feasibility Trial of a Legal Navigation Program to Address Cancer-related Legal Barriers
Brief Title: Legal Evaluation for Greater Access to Cancer Care (LEGAL-CARE)
Acronym: LEGAL-CARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Triage Cancer (Unknown)
Responsible Party: Principal Investigator, Qasim Hussaini, Assistant Professor of Medicine, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 300014052; UAB O'Neal Invest Award (Other Grant/Funding Number: University of Alabama at Birmingham Comprehensive Cancer Center)
Record Dates: First submitted 2025-09-03; First posted 2025-09-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Cancer
Keywords: legal; navigation; legal barriers; cancer; oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Legal Intervention Arm (Experimental): There will be 6 proactive legal intervention cycles. During each, an attorney will proactively reach out to the patient or caregiver via telephone or video call within the first month of enrollment to identify and address legal barriers in areas such as health insurance, financial, disability insurance, employment, and other (estate planning, advanced directives, life insurance, family law). The attorney will guide patients and caregivers through necessary actions, and provide resolution. Baseline, 3, and 6 months surveys will be collected, as well as additional surveys at the 1, 2, 3, 4, 5, and 6 month check ins with the legal team.
  Interventions: Behavioral: Legal Navigation

INTERVENTIONS:
Behavioral: Legal Navigation — • Participants will receive monthly outreach from a trained legal navigator over a 6-month period. The legal navigator is a lawyer (Juris Doctor, or JD) who will proactively address specific legal barriers the patient may encounter during treatment. Communication will include phone calls (and if requested, virtual consultations) tailored to patient needs. In between legal outreach periods, patients may call the legal navigator team themselves for legal needs that may arise.
  Other Names: Navigation

SUMMARY:
This study aims to help patients with cancer facing legal issues. The investigators noticed that many patients struggle with laws and regulations related to disability benefits, employment rules, health insurance denials, and financial assistance barriers among many others. To understand this better, the investigators conducted the first nationwide study on how legal problems affect patients with cancer. Investigators noted a striking prevalence of legal issues in patients with cancer - most struggled with 2 or more legal issues that impacted their care. These legal issues looked different for those with different socioeconomic backgrounds. In a second study, the investigators also found healthcare workers (HCWs) including social workers and navigators feel underprepared to counsel patients on legal topics.

Now, the investigators launching a pilot program called LEGAL-CARE at the O'Neal Comprehensive Cancer Center at the University of Alabama at Birmingham (UAB) to help patients navigate these legal hurdles. Patients in the study will receive legal navigation, where they will get help with legal issues related to their cancer treatment.

The investigators will look at how practical or feasible such a program is, and how it affects patients' lives over time. The investigators will check in with the participants at regular time intervals to see if they feel less stressed about money, have a better quality of life, and use healthcare services differently. The investigators will also see if the program helps reduce the number of legal problems they face. Finally, the investigators will discuss with the participants about how this legal intervention could be made better.

This study is important because it's the first of its kind. It will give insights into how legal problems impact patients with cancer and how addressing these issues can improve their lives. Plus, it'll help the investigators better understand implementing similar programs in other places. Overall, it's a partnership between O'Neal, national legal assistance organizations, and the Birmingham community to make life easier for people dealing with cancer and legal challenges. Ultimately, the goal will be to take what the investigators learn here to run a larger multi-site trial.

DETAILED DESCRIPTION:
Despite an adept social and navigation workforce, the regulatory and legal landscape for patients with cancer has become increasingly difficult to navigate. Many barriers faced by patients are entrenched in local, state, and federal policies that require expertise in both social needs and the law. Recently, the investigators led the first nationwide study investigating the extent to which patients with cancer encounter legal barriers related to disability, employment, health insurance, and financial assistance. There is an urgent need for evidence on how interventions can mitigate cancer-related legal barriers and impact care.

The Legal Evaluation for Greater Access to Cancer Care (LEGAL-CARE) is a pilot feasibility trial of a legal navigation program to address cancer-related legal barriers. A small cohort of patients will be offered at least one cycle of legal intervention over a 6-month period. Legal intervention is defined as a legal navigator proactively reaching out to the patient to discuss legal hardship during their treatment. This study will take place in the medical oncology clinics at the O'Neal Comprehensive Cancer Center. Inclusion criteria includes any adult aged 18 or older with a new diagnosis of advanced stage cancer (stages III or IV) requiring systemic therapy that is being seen in clinic. The objectives of this study are to evaluate the feasibility of a legal intervention, and understand patient perceptions utilizing semi-structured interviews. Additionally, it will assess patient-reported financial toxicity, quality of life, and health care utilization between patients receiving legal navigation. The investigators hypothesize this legal intervention would be feasible, acceptable and implemented as intended by the research protocol, while also demonstrating measurable improvement in patient outcomes.

The LEGAL-CARE study is relevant to the investigators' catchment area with a unique legal and regulatory landscape in Alabama, and situated in the context of recent American Society of Clinical Oncology (ASCO)-level and federal-level policy developments examining the role of legal services and SDOH in the context of cancer care. This study is significant as it will be the first to prospectively investigate the impact of legal barriers on patient care. It is innovative for multiple reasons. It employs a unique legal intervention and assesses the feasibility and acceptability of the intervention in preparation for a larger multi-site trial. It leverages a unique partnership between O'Neal's social work service, and the nation's largest organization providing legal assistance to patients with cancer, and community legal aid organizations in Birmingham. Finally, it results in a rich mixed methods analytic dataset that will allow implementation-related information from the intervention to be utilized in an R01 grant to scale this regionally.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria includes adults ≥18 years old
* New de novo advanced stage cancer (stages III/IV) requiring systemic therapy..

Exclusion Criteria:

* non-melanoma skin cancer
* benign cancer or in-situ tumor
* a recurrence of a previously diagnosed cancer
* a hospice encounter in the past year
* those unable to complete surveys
* unable to communicate fluently in English
* unable to provide consent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility Benchmarks | 6 months
  Feasibility will be measured by
  1. retention of ≥70% of enrolled patients at 6 months and
  2. ≥75% completion of biweekly surveys among retained patients.
  Acceptability will be measured by the Acceptability of Intervention Measure (AIM), 4 items on a 5-point Likert scale (1-5; higher = more acceptable).
  Appropriateness will be measured by the Intervention Appropriateness Measure (IAM), 4 items on a 5-point Likert scale (1-5; higher = more appropriate).
  Feasibility (perceptions) will be measured by the Feasibility of Intervention Measure (FIM), 4 items on a 5-point Likert scale (1-5; higher = more feasible).

SECONDARY OUTCOMES:
Patient perceptions of legal intervention impact | At the end of 6 month legal intervention
  Using semi-structured interviews, we will explore the effects of legal intervention on (1) legal barriers encountered during care, (2) perceived change in quality of life, (3) recommendations for modifying delivery intervention including dose, frequency, duration and content, and (4) current retention and future participation in clinical trials
Financial hardship, health-related quality of life, legal burden, administrative burden, and health care utilization | 6 months
  Financial toxicity measured by the Comprehensive Score for Financial Toxicity (COST-FACIT), range 0-44 with lower scores indicating worse toxicity.
  Health-related quality of life measured by the Functional Assessment of Cancer Therapy - General (FACT-G), range 0-108 with higher scores indicating better quality of life.
  Legal burden assessed by an investigator-developed questionnaire, with higher scores indicating greater burden.
  Administrative burden assessed by an investigator-developed questionnaire, with higher scores indicating greater burden.
  Health care utilization assessed from electronic medical record review, including emergency department visits, hospitalizations, intensive care admissions, urgent care visits, palliative care use, and treatment delays, reported as counts per patient at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Qasim M Hussaini, MD, MS, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The Kirklin Clinic, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided
Consideration will be given to sharing of IDP as the study progresses.

DOCUMENTS (1):
  • Study Protocol (2025-02-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT07197515/Prot_000.pdf